CLINICAL TRIAL: NCT01482949
Title: A Rollover Phase II Study Testing the Biologic Activity and Safety of AGS-003 in Renal Cell Carcinoma Subjects With Prolonged Response or Stable Disease and Ongoing AGS-003 Treatment in Protocol AGS-003-004 or AGS-003-006
Brief Title: A Rollover Protocol for Subjects Previously Treated With AGS-003
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Argos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGS-003-005
Record Dates: First submitted 2011-11-17; First posted 2011-12-01 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Renal Cell Carcinoma
Keywords: RCC; Kidney Cancer; Renal Cancer; Arcelis
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AGS-003 in combination with sunitinib (Experimental): Subjects will undergo Induction (AGS-003 every 3 weeks until 5 doses are administered) followed by Booster (AGS-003 at 3 month intervals). Subjects that will begin sunitinib therapy will be on this arm.
  Interventions: Drug: AGS-003

INTERVENTIONS:
Drug: AGS-003 — Autologous Dendritic Cell Immunotherapy
  Other Names: Arcelis

SUMMARY:
The purpose of this study is to evaluate clinical response to AGS-003 alone or in combination with sunitinib therapy.

DETAILED DESCRIPTION:
AGS-003-005 is a rollover, open label, Phase II clinical study testing the biologic activity and safety of AGS-003 in subjects who have experienced either partial responses or prolonged stable disease and continue to benefit from ongoing treatment with AGS-003 in protocols AGS-003-004 or AGS-003-006.

Rollover subjects from AGS-003-004 will continue with AGS-003 monotherapy booster dosing until disease progression or until a discontinuation criterion is reached.

Subjects that progress on AGS-003 monotherapy (from the AGS-003-004 protocol) may start sunitinib treatment and re-initiate AGS-003 therapy beginning with the induction phase dosing schedule.

Rollover subjects from AGS-003-006 will continue sunitinib dosing in combination with booster dosing of AGS-003 until disease progression or until a discontinuation criterion is reached.

If a subject has disease progression due to a new tumor lesion, upon consultation between the investigator, Argos representatives and the Argos medical monitor, the subject may be considered for re-manufacture of study product (from the new metastatic lesion) and dosing with this new product in combination with sunitinib beginning with the induction phase dosing schedule.

For those subjects initiating treatment with the induction phase as described above, restaging imaging occurs at screening (baseline), prior to the fifth dose in the induction phase (as applicable) and every 12 weeks during the booster phase (at the start of the sunitinib holiday, 2 weeks prior to the next AGS-003 dose).

For subjects on combination therapy, if dosing with sunitinib is stopped due to sunitinib-related issues, treatment with AGS-003 may continue.

Close-out visits will occur upon disease progression (other than circumstances discussed above which are eligible for re-induction) or upon decision to terminate the study by the sponsor.

Quarterly follow-up for survival for each subject will occur by telephone interview for 1 year following the last AGS-003 administration or study termination.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Subjects are receiving ongoing treatment with AGS-003 in protocol AGS- 003-004 or AGS-003-006.
* Measurable disease that can be monitored per RECIST throughout the course of study participation.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematologic function, as defined by the following criteria:

  1. White blood cell (WBC) ≥ 4000/µL (≥ 4.0 x 103/µL)
  2. Absolute neutrophil count (ANC) ≥ 1500/µL (≥ 1.5 x 103/µL)
  3. Platelets ≥ 100,000/µL (≥ 100 x 103/µL)
  4. Hemoglobin (Hgb) ≥ 9.0 g/dL
* Adequate renal and hepatic function, as defined by the following criteria:

  1. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or, if serum creatinine > 1.5 x ULN, estimated glomerular filtration rate (eGFR) ≥ 30 mL/min
  2. Total serum bilirubin ≤ 1.5 x ULN
  3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN, or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy
* Adequate coagulation function as defined by the following criteria:

  1. Prothrombin time (PT) ≤ 1.5 x ULN
  2. Activated partial thromboplastin time (PTT) < 1.5 x ULN
  3. Corrected calcium ≤ 11.5 mg/dL
* Negative serum pregnancy test for female subjects with reproductive potential, and agreement of all male and female subjects of reproductive potential to use a reliable form of contraception during the study and for 12 weeks after the last dose of study drug
* Able to abstain from taking prohibited drugs, either prescription or non- prescription, during the treatment phase of the study
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment
* No brain metastases detected by magnetic resonance imaging (MRI).

Exclusion Criteria:

* Any serious medical condition considered by the investigator to constitute an unwarranted high risk for investigational treatment
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or evidence of brain or leptomeningeal disease on screening computed tomography (CT) scan or MRI
* Pregnancy or breastfeeding
* Active autoimmune disease or condition requiring chronic immunosuppressive therapy

NOTE: Abnormal laboratory values for autoimmunity markers in the absence of other signs/symptoms of autoimmune disease are not exclusionary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-09; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Tumor response | From date of registration until either disease progression, meeting a discontinuation criterion, or death; assessed up to 36 months.
  Clinical antitumor activity of AGS-003 will be assessed as an objective tumor response by Response Evaluation Criteria in Solid Tumors (RECIST).

SECONDARY OUTCOMES:
Clinical benefit (stable disease or response) | From date of registration until either disease progression, meeting a discontinuation criterion, or death; assessed up to 36 months.
  Clinical benefit measured as Stable Disease (SD), Partial Response (PR), and Complete Response (CR) rate to the treatment regimen. Tumor response is verified using standard definitions of RECIST
Immune function | From date of registration until either disease progression, meeting a discontinuation criterion, or death; assessed up to 36 months.
  Analyses of immune function will be performed. This will include, but not limited to, assessment of T cell and antigen presenting cell populations, including effector memory, cytotoxic lymphocytes (CTLs), and regulatory T cells. Blood and plasma specimens for these analyses will be collected at specified time points and is optional for subjects continuing with booster treatments.
Progression Free Survival (PFS) | From date of registration until either disease progression, meeting a discontinuation criterion, or death; assessed up to 36 months.
  Evaluate PFS from the date of registration until PFS is reached per RECIST
Overall Survival (OS) | From date of registration until either disease progression, meeting a discontinuation criterion, or death; assessed up to 36 months.
  Evaluate OS from date of registration until date of death.
Treatment-emergent Adverse Events | From date of registration until either disease progression, meeting a discontinuation criterion, or death; assessed up to 36 months.
  Monitor incidence of treatment-emergent Adverse Events.
Monitor clinical chemistry, hematology, and urinalysis for treatment-emergent changes from baseline | From date of registration until either disease progression, meeting a discontinuation criterion, or death; assessed up to 36 months.
  Clinical laboratory values will be monitored for changes from baseline.
Physical Examinations | From date of registration until either disease progression, meeting a discontinuation criterion, or death; assessed up to 36 months.
  Monitor changes from baseline in physical examinations
Vital Signs | From date of registration until either disease progression, meeting a discontinuation criterion, or death; assessed up to 36 months.
  Monitor changes from baseline in vital signs
Monitor signs and symptoms indicating treatment-emergent autoimmunity | From date of registration until either disease progression, meeting a discontinuation criterion, or death; assessed up to 36 months.
  Autoimmunity evaluations will be measured by clinical signs and symptoms (e.g., rash, cytopenias, and arthralgias) and by laboratory assessments. These assessments will be monitored as long as the subject is receiving AGS-003.
Monitor for lymph node adenopathy | From date of registration until either disease progression, meeting a discontinuation criterion, or death; assessed up to 36 months.
  The draining lymph nodes (axillary and inguinal) will be evaluated for changes from baseline in size, tenderness, or inflammation. These assessments will be monitored as long as the subject is receiving AGS-003.
Injection Site Reaction | From date of registration until either disease progression, meeting a discontinuation criterion, or death; assessed up to 36 months.
  Monitor changes from baseline in injection site reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Lee F Allen, M.D., Ph.D., Study Director — Argos Therapeutics
Locations (1):
- University of Minnesota Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No